CLINICAL TRIAL: NCT04692090
Title: Effects of Yoga on Phase Angle and Quality of Life in Patients With Breast Cancer: A Randomized, Single-blind, Controlled Trial
Brief Title: Effects of Yoga on Phase Angle and Quality of Life in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sibel Eyigor, Professor in Ege University Faculty of Medicine, Physical Medicine and Rehabilitation Department, Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yoga-PA
Record Dates: First submitted 2020-12-30; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
Keywords: Phase Angle; Hatha Yoga; Breast Cancer; Quality of Life
MeSH Terms: conditions — Breast Neoplasms | interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga Group (Experimental): Hatha yoga will be practiced twice a week for 10 weeks
  Interventions: Other: Yoga
- Control group (No Intervention): This group will not have any intervention.

INTERVENTIONS:
Other: Yoga — Each class started with a check-in period during which any questions or concerns could be raised, after which the patients were given 5 minutes for seated meditation and 10 minutes for Shavasana (lying down in a restorative position).
  The following poses were instructed during the course: standing poses with mountain pose (tadasana), chair pose (utkatasana), extended triangle pose (utthita trikonasana), extended side angle pose (utthita parshvakonasana), warrior 1 (virabhadrasana 1), warrior 2 (virabhadrasana 2) and tree pose (vrikshasana). The intervention was applied twice a week for 10 weeks.
  Arms: Yoga Group

SUMMARY:
In this study,we aimed to examine the effects of Hatha yoga on PA and QoL in patients with breast cancer.

Patients will be randomized to receive the yoga group and the control group.Hatha yoga will be practiced twice a week for 10 weeks for intervention group.The PA of the patients will be assessed using a body analysis instrument and QoL was evaluated with an EORTC-Q questionnaire both before treatment and at week 10.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 70, witha diagnosis of breast cancer

Exclusion Criteria:

* Patients with recurrent or progressive disease, or with serious heart or pulmonary disease, with uncontrolled hypertension, infection, cognitive function disorder, psychiatric disease or musculoskeletal system conditions that would prevent exercise, and those who had taken part in a regular exercise program

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2015-11-05 (Actual); Study Completion 2015-11-05 (Actual)

PRIMARY OUTCOMES:
Phase Angle | 10 weeks
  Phase angle was evaluated with a Tanita body composition monitor (Tanita Corp., Tokyo, Japan). Electrodes are placed on both feet and both hands that send electrical signals from the body to a single independent unit. Voltages are measured at the top of the thumbs on both hands and both heels. A high-frequency electric current (90μA at 50 kHz) is applied, and the Resistance (R) and Reactance (xc) values are measured between the hands and feet. Internal software calculates the phase angle based on the following formula: Phase angle (PhA) = Reactance (xc) / Resistance (R) * (180 / π)

SECONDARY OUTCOMES:
The European Organization for Research and Treatment of Cancer Quality of life (EORTC QLQ-C30) questionnaire | 10 weeks
  The European Organization for Research and Treatment of Cancer Quality of life (EORTC QLQ-C30) questionnaire; This 30-question survey is conducted to evaluate QoL in patients with breast cancer and assesses any symptoms that occurred in the previous two weeks. The questionnaires are divided into three scales: global health scale (GHS), functional scale (FS), and symptom scale (SS). High scores in the functional and global health scales indicate a good QoL, while high scores on the symptom scale point to a high level of problems
Arm Volume | 10 weeks
  Patients were also evaluated for the lymphedema of the limbs is assessed through circumferential and volumetric methods. Circumferential upper limb measurements were carried out with the arm abducted to 30°, starting at the level of the carpometacarpal joint, and at every 5 cm proximal to this point along with both limbs
Body-Mass Index | 10 weeks
  Body Mass Index is a simple calculation using a person's height and weight. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.

IPD SHARING:
Plan to Share IPD: No